CLINICAL TRIAL: NCT03277378
Title: Randomized, Controlled, Single Blind, Prospective, Multicenter Study Evaluating Anatomic Versus Targeted Lead Placement for BurstDR Therapy During the Trial Evaluation Period. (DELIVERY)
Brief Title: Evaluating Anatomic Versus Targeted Lead Placement for Burst Stimulation Therapy During the Trial
Acronym: DELIVERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJM-CIP-10116
Record Dates: First submitted 2017-09-04; First posted 2017-09-11 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Chronic, Intractable Pain of the Trunk and/or Lower Limbs
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Group 1 (AB) (Active Comparator): Group 1 (AB): anatomic lead placement followed by BurstDR™ stimulation during an initial trial evaluation period
  Interventions: Device: lead placement followed by BurstDR stimulation
- Group 2 (TB) (Active Comparator): Group 2 (TB): targeted lead placement followed by BurstDR™ stimulation during an initial trial evaluation period
  Interventions: Device: lead placement followed by BurstDR stimulation

INTERVENTIONS:
Device: lead placement followed by BurstDR stimulation — lead placement followed by BurstDR stimulation
  Other Names: Spinal Cord Stimulation non-surgical Leads; Spinal Cord Stimulation Clinician Programmer; Spinal Cord Stimulation Patient Controller

SUMMARY:
Prospective, multi-center, randomized, single blind study

DETAILED DESCRIPTION:
This clinical investigation compares success rates for anatomically placed leads to conventional, targeted lead placement for BurstDR™ during the trial evaluation period with the St Jude Medical™ Invisible Trial System. Subjects will be blinded to treatment group and randomized in a 1:1 ratio as follows:

Group 1 (AB): anatomic lead placement followed by BurstDR™ stimulation during an initial trial evaluation period Group 2 (TB): targeted lead placement followed by BurstDR™ stimulation during an initial trial evaluation period

If the subject qualifies for permanent system implant according to pre-defined criteria after the initial trial evaluation period, the subject will exit the clinical investigation and continue their treatment per the physician's standard of care. Subjects who do not qualify for permanent system implant according to pre-defined criteria after the initial trial evaluation period may participate in an extended trial evaluation period, per physician discretion, during which they will be programmed with tonic stimulation. Subjects continuing to an extended trial evaluation period will be followed through the completion of the extended trial period. At the end of the extended trial evaluation period, subjects will exit the clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient indicated for Spinal Cord Stimulation therapy in accordance with the approved labeling.
2. Patient's pain profile indicates appropriate lead placement would be at one or more levels from T7 to T10, to achieve pain coverage.
3. Patient has a baseline score on the Numerical Rating Scale ≥6 over the past 24 hours for 'average overall pain'specific to the area(s) of chronic pain that will be treated with spinal cord stimulation.
4. Patient is considered by the Study Investigator as a candidate for implantation of a spinal cord stimulator system according to the system Instructions for Use.
5. Patient is >18 years of age at the time of enrollment.
6. Patient is willing to adhere to the study requirements, including compliance with and completion of all study visits.
7. Patient has signed and received a copy of the Ethical Committee/Independent Review Board approved informed consent.

Exclusion Criteria:

1. Patient currently has a spinal cord stimulation system implanted.
2. Patient has previously failed a spinal cord stimulation therapy (either trial system evaluation or permanent system implant).
3. Patient has a primary diagnosis of Peripheral Vascular Disease (PVD), Angina Pectoris, or Chronic Migraine.
4. Patient is scheduled to undergo an on-the-table trial evaluation (aka all-in-one procedure)
5. Patient is scheduled to be implanted with (a) surgical paddle trial lead(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Capobianco, PhD, Study Director — Abbott
Locations (25):
- United States (13):
  - Jason Edward Pope, MD, Santa Rosa, California
  - Comprehensive Spine Institute, Clearwater, Florida
  - Florida Pain Institute, Merritt Island, Florida
  - National Pain Institute Winter Park, Winter Park, Florida
  - Rush University, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Advanced Pain Care, Las Vegas, Nevada
  - Nevada Advanced Pain Specialists, Reno, Nevada
  - Oregon Health & Science University, Portland, Oregon
  - Spinal Diagnostics, Tualatin, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Precision Spine Care, Tyler, Texas
  - St. Mary's Hospital, Huntington, West Virginia
- Australia (2):
  - Frankston Pain Management, Frankston
  - North Shore Private Hospital, Saint Leonards
- Austria (2):
  - Hospital Elisabethinen GmbH, Graz
  - Wilhelminenspital Wien, Vienna
- Germany (4):
  - Sana Kliniken Duisburg Gm.bH, Duisburg
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf
  - Hospital Gera -Zentrum für interdisziplinäre Schmerztherapie, Gera
  - Klinikum Nürnberg Sud, Nuremberg
- Fondazione Salvatore Maugeri, Pavia, Italy
- Netherlands (2):
  - Alrijne Ziekenhuis, Leiderdorp
  - Stichting Rijnstate Ziekenhuis - Velp, Velp
- University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject enrollment for the DELIVERY study began on 22 September 2017, at 23 clinical sites in the United States, Europe, and Australia. A total of 270 subjects were randomized into the two treatment groups (Anatomic Lead Placement and Targeted lead placement).
Pre-assignment Details: A total of 288 subjects were screened, of which 18 subjects were withdrawn before randomization due to unmet inclusion/exclusion criteria (n=6), withdrawal of the consent (n=11) and subject was on the clinic's wait list to receive an implant only after the study closed (n=1). The last follow-up visit occurred on 27 August 2018.
Period: Overall Study
Arm/Group | Group 1 (AB) | Group 2 (TB)
Started | 135 | 135
Received Lead Implant | 129 | 123
Completed Initial Trial | 126 | 122
Qualified for Permanent Implant | 103 | 93
Not Qualified for Permanent Implant | 19 | 20
Completed Extended Trial With Tonic Stim | 8 | 12
Exit Study | 11 | 8
Completed | 111 | 101
Not Completed | 24 | 34

BASELINE CHARACTERISTICS:
Population: The baseline characteristics for all subjects randomized to anatomic or targeted lead placement were measured.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (AB) | Group 2 (TB) | Total
Number analyzed (Participants) | 135 | 135 | 270
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.8 (13.2) | 63.9 (13.8) | 62.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 87 | 165
  Male | 57 | 48 | 105
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of participants analyzed includes subjects who were available at that time of analysis
  Participants
    number analyzed (Participants) | 116 | 116 | 232
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Black or African American | 5 | 3 | 8
    White | 103 | 98 | 201
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 7 | 14 | 21
Region of Enrollment [Number; unit: participants]
  Austria | 2 | 3 | 5
  Netherlands | 1 | 1 | 2
  Italy | 4 | 4 | 8
  Australia | 7 | 7 | 14
  Germany | 12 | 11 | 23
  United States | 109 | 109 | 218
Years of having chronic pain [Mean (Standard Deviation); unit: years] | 12.23 (11.83) | 10.69 (11.11) | 11.46 (11.48)

OUTCOME MEASURES:

1. Primary Outcome: Qualification Rate for Permanent System Implant at the End of the Initial Trial Evaluation Period
Description: The primary endpoint is the qualification rate for permanent system implant at the end of the initial trial evaluation period.
  Qualification for permanent system implant was defined by a composite where all the following conditions were met:
  * ≥ 50% patient reported pain relief (PRP) at the end of the trial evaluation
  * Trial evaluation period lasted for a minimum of 3 days
  * Physician recommends subject for permanent system implant
  * Subject reports a willingness to pursue a permanent system implant
  Subjects did not qualify for permanent system implant if they met both of the following:
  * < 50% PRP (patient reported pain relief) at the end of the trial evaluation
  * Trial evaluation period lasted for a minimum of 5 days
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 122 | 113
Participants | 103 | 93
Statistical Analysis 1: Comparison: Group 1 (AB) vs Group 2 (TB); The hypothesis was formally addressed as: H0: AB - TB ≤ -15% H1: AB - TB > -15% where AB = permanent system qualification rate of Group 1 (AB) TB = permanent system qualification rate of Group 2 (TB); Test type: Non-Inferiority — The hypothesis was tested at the 5% significance level; p = 0.0003, Farrington- Manning non-inferioirty test

2. Secondary Outcome: Rate of Physician Preference for Anatomic Placement Versus Targeted Placement at the End of the Study
Description: The physician preference for placement of leads was noted by giving them the option of choosing which lead placement technique they preferred - anatomic or targeted lead placement technique.
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The analysis population included physicians who had performed both types of lead placement procedures.
Measure: Count of Participants; unit: Participants
Groups:
- Physicians Who Prefer Anatomic Lead Placement: Physicians who preferred anatomic placement of leads
- Physicians Who Prefer Targeted Placement of Leads: Physicians who prefered targeted placement of leads
Arm/Group | Physicians Who Prefer Anatomic Lead Placement | Physicians Who Prefer Targeted Placement of Leads
Number analyzed (Participants) | 20 | 20
Participants | 14 | 6
Statistical Analysis 1: Comparison: Physicians Who Prefer Anatomic Lead Placement vs Physicians Who Prefer Targeted Placement of Leads; The hypothesis was formally addressed as: H0: P ≤ 60% H1: P > 60% where P= percentage of physician prefer anatomic placement over targeted placement. The analysis population included physicians who have performed both placement procedures. The hypothesis was tested at the 5% significance level; Test type: Other; p = 0.2500, Chi-squared

3. Other Pre Specified Outcome: Procedural Characteristics of Subjects With One Trial Lead Implanted (US)
Description: Procedural characteristics including overall procedure time (room-in to room-out, implant procedure time (needle-in to needle-out, and the intraoperative time for the fluoroscopy procedure were measured.
Time Frame: Trial system implant
Population: Subjects include those who had one trial lead implanted in sites in the United States.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 4 | 7
Minutes
  Overall procedure time | 57.3 (4.7) | 52.9 (16.9)
  Implant procedure time | 38 (9.4) | 30.3 (14.2)
  Intraoperative fluoroscopy time | 2.48 (1.95) | 2.65 (2.05)

4. Other Pre Specified Outcome: Procedural Characteristics of Subjects With One Trial Lead Implanted (OUS)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had one trial lead implanted in sites outside the United States.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 7 | 6
Minutes
  Overall procedure time | 38 (11.8) | 46.2 (19.2)
  Implant procedure time | 11.6 (6.8) | 21.5 (15.5)
  Intraoperative fluoroscopy time | 4.22 (2.56) | 4.28 (2.68)

5. Other Pre Specified Outcome: Procedural Characteristics of Subjects With One Trial Lead Implanted (Worldwide)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had one trial lead implanted in sites worldwide
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 11 | 13
Minutes
  Overall procedure time | 45.0 (13.6) | 49.8 (17.6)
  Implant procedure time | 21.2 (15.2) | 26.2 (14.9)
  Intraoperative fluoroscopy time | 3.59 (2.42) | 3.40 (2.41)

6. Other Pre Specified Outcome: Procedural Characteristics of Subjects With Two Trial Leads Implanted (US)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had two trial leads implanted in sites in the United States.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 99 | 90
Minutes
  Overall procedure time | 40 (12.4) | 45 (13.7)
  Implant procedure time | 14 (8.2) | 19.9 (10)
  Intraoperative fluoroscopy time | 1.52 (0.98) | 1.68 (1.24)

7. Other Pre Specified Outcome: Procedural Characteristics of Subjects With Two Trial Leads Implanted (OUS)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had two trial leads implanted in sites outside the United States.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 7 | 7
Minutes
  Overall procedure time | 45.9 (10.4) | 57.3 (15.8)
  Implant procedure time | 19.1 (11.7) | 30 (14.2)
  Intraoperative fluoroscopy time | 3.5 (1.56) | 3.24 (1.24)

8. Other Pre Specified Outcome: Procedural Characteristics of Subjects With Two Trial Leads Implanted (Worldwide)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had two trial leads implanted in sites worldwide
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 106 | 97
Minutes
  Overall procedure time | 40.4 (12.3) | 45.9 (14.1)
  Implant procedure time | 14.3 (8.5) | 20.6 (10.6)
  Intraoperative fluoroscopy time | 1.65 (1.13) | 1.79 (1.30)

9. Other Pre Specified Outcome: Procedural Characteristics of Subjects With One Permanent Lead Implanted (OUS)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had one permanent lead implanted in sites outside the United States.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 9 | 10
Minutes
  Overall procedure time | 59.6 (16.2) | 68.6 (19.7)
  Implant procedure time | 11.6 (9.4) | 22.6 (12.2)
  Intraoperative fluoroscopy time | 2.12 (0.88) | 2.83 (1.64)

10. Other Pre Specified Outcome: Procedural Characteristics of Subjects With Two Permanent Leads Implanted (OUS)
Description: as for outcome 3
Time Frame: Trial system implant
Population: Subjects include those who had two permanent leads implanted in sites outside the United States.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 3 | 3
Minutes
  Overall procedure time | 56 (4.6) | 92.3 (23.7)
  Implant procedure time | 19.3 (5.1) | 27.3 (6.5)
  Intraoperative fluoroscopy time | 5.96 (3.09) | 4.93 (4.45)

11. Other Pre Specified Outcome: Programming Time Needed for Each Randomized Group
Description: The programming time observed for both randomized groups
Time Frame: Trial system implant
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 127 | 123
Minutes | 5 (6.4) | 6 (6)

12. Other Pre Specified Outcome: Change From Pre-implant Numerical Rating Scale (NRS) in Each Randomized Group to End of Initial Trial Evaluation Period
Description: Subjects were interviewed using the pain NRS scale consisting of 1 question and were asked to rate their average pain specific to the area(s) of chronic pain being treated over the past 24 hours on a 0 (no pain) to 10 (worst imaginable pain) scale. A higher score indicates a higher pain level.
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 124 | 121
Score on a scale | 4.2 (2.8) | 4.3 (2.7)

13. Other Pre Specified Outcome: Change From Pre-implant Numerical Rating Scale (NRS) in Each Randomized Group to the End of the Extended Trial Evaluation Period
Description: as for outcome 12
Time Frame: From pre-implant to end of extended trial period, a minimum of 5 days BurstDR stimulation plus an additional minimum of 3 days tonic stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 10 | 14
Score on a scale | 2.4 (2.6) | 2.6 (2.2)

14. Other Pre Specified Outcome: Number of Subjects Who Have Affirmative Assessment for Each of the Independent Criteria Required for Qualification for Permanent Implant
Description: Number of subjects in each randomized group who have affirmative assessment for each of the independent criteria required for qualification for permanent implant
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 126 | 122
Participants
  ≥ 50% patient reported pain relief (PRP) | 107 | 99
  Trial period lasted for a minimum of 3 days | 126 | 122
  Physician recommendation for permanent implant | 109 | 104
  Subject's willingness for a permanent implant | 106 | 100

15. Other Pre Specified Outcome: Proportion of Subjects Who do Not Qualify for Permanent Implant But Proceeded With Permanent Implant Per Physician Discretion.
Description: Number of subjects in each randomized group who do not qualify for permanent implant but proceeded with permanent implant per physician discretion.
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 126 | 122
Participants | 1 | 2

16. Other Pre Specified Outcome: Time From Trial System to ≥ 50% Patient Reported Pain Relief (PRP)
Description: Time from trial system to ≥ 50% patient reported pain relief measured by the number of days (also known as " wash-in period")
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 64 | 61
Days | 3.0 (2.0) | 3.3 (2.8)

17. Other Pre Specified Outcome: Rate of Serious Adverse Device Effects (SADE) Based on Randomization
Description: Rate of serious adverse device effects based on each randomized group.
Time Frame: From pre-implant to exit of the study, approximately 3 to 14 days
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 135 | 135
Participants | 1 | 1

18. Other Pre Specified Outcome: Number and Proportion of Meaningful Lead Migrations During the Initial Trial Evaluation Periods by Treatment Group
Description: A meaningful lead migration is defined as a lead migration resulting in the inability to program for therapeutic response
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 129 | 123
Participants | 1 | 1

19. Other Pre Specified Outcome: Number and Proportion of Meaningful Lead Migrations During Initial Trial Evaluation Period by Lead Type
Description: The number and proportion of meaningful lead migrations during initial trial evaluation period was assessed based on lead type (either Temporary Lead Implant or Permanent Lead Implant). A meaningful lead migration is defined as a lead migration resulting in the inability to program for therapeutic response
Time Frame: From pre-implant to end of initial trial evaluation period, 3 to 5 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Groups:
- Subjects With Temporary Lead Implant: Subjects who had temporary lead implant after randomization
- Subjects With Permanent Lead Implant: Subjects who had Permanent lead implant after randomization
Arm/Group | Subjects With Temporary Lead Implant | Subjects With Permanent Lead Implant
Number analyzed (Participants) | 227 | 25
Participants | 2 | 0

20. Other Pre Specified Outcome: Clinician Assessment of Anesthesia Related Difficulty and Lead Placement Difficulty
Description: Clinician assessment of anesthesia related difficulty and lead placement difficulty using a Likert scale ranging from ' No difficulty' to extreme difficulty and clinician affinity for lead placement technique at the end of the trial implant procedure.
Time Frame: Trial system implant
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 129 | 123
Participants
  Anesthesia related difficulty: No difficulty | 113 | 99
  Anesthesia related difficulty: Little difficulty | 12 | 17
  Anesthesia related difficulty: Moderate difficulty | 4 | 7
  Anesthesia related difficulty: Severe difficulty | 0 | 0
  Anesthesia related difficulty: Extreme difficulty | 0 | 0
  Anesthesia related difficulty: Could not place leads | 0 | 0
  Lead placement difficulty: No difficulty | 82 | 77
  Lead placement difficulty: Little difficulty | 28 | 28
  Lead placement difficulty: Moderate difficulty | 14 | 16
  Lead placement difficulty: Severe difficulty | 1 | 1
  Lead placement difficulty: Extreme difficulty | 2 | 0
  Lead placement difficulty: Could not place leads | 2 | 1

21. Other Pre Specified Outcome: Clinician Affinity for Lead Placement Technique at the End of Trial Procedure
Description: Clinician affinity for lead placement technique at the end of the trial implant procedure using a Likert scale ranging from 0 being 'Not all' to 4 being ' very much'.
Time Frame: Trial system implant
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 129 | 123
Participants
  0 | 4 | 1
  1 | 3 | 3
  2 | 4 | 3
  3 | 13 | 4
  4 | 46 | 11
  This was my usual practice | 59 | 101

22. Other Pre Specified Outcome: Permanent System Qualification Rate at the End of Extended Trial Period
Description: The qualification rate for permanent implant was calculated for the subjects who completed the extended trial period.
Time Frame: as for outcome 13
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 (AB) | Group 2 (TB)
Number analyzed (Participants) | 10 | 14
Participants | 5 | 11

ADVERSE EVENTS:
Time Frame: Approximately 3 to 14 days
Arm/Group | Group 1 (AB) | Group 2 (TB)
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/135
Serious Adverse Events (participants affected / at risk) | 2/135 | 1/135
Other Adverse Events (participants affected / at risk) | 4/135 | 6/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (AB) (N=135) | Group 2 (TB) (N=135)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Spinal Cord Compression (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stimulation in unwanted places (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (AB) (N=135) | Group 2 (TB) (N=135)
Hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lead Migration (Product Issues) | 2 (2) | 2 (2)
Unpleasant sensations or Motor disturbances Including Involuntary Movement caused by high output (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Persistant pain lead site (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cerebrospinal fluid leakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
New leg pain on walking instead of original dysaesthetic sensation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was designed to collect data during the initial trial period only. Anatomic placement of leads may not provide adequate paresthesia coverage for patients wishing to periodically use a paresthesia-based stimulation design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03277378/Prot_SAP_000.pdf